CLINICAL TRIAL: NCT04876235
Title: Efficacy and Safety of Double-pigtail Plastic Versus Lumen-apposing Metal Stents for Transmural Drainage of Walled-off Necrosis
Brief Title: A Comparison Between Lumen-apposing Metal Stent and Double-pigtail Plastic Stents for Treatment of Walled-off Necrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Deputy irector, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-03-221
Record Dates: First submitted 2021-04-30; First posted 2021-05-06 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Walled-off Necrosis
Keywords: endoscopic ultrasound guided drainage; Lumen-apposing metal stent; double-pigtail plastic stents; Walled-off necrosis
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAMS group (Experimental): place LAMS under endoscopic ultrasound. Direct endoscopic necrosectomy(DEN) was performed through the LAMS with a forward viewing gastroscope if necessary
  Interventions: Procedure: endoscopic ultrasound; Device: lumen-apposing metal stent
- DPPS group (Active Comparator): Place DPPS under endoscopic ultrasound. When required, DEN was performed once the cystogastrostomy/duodenostomy tract had matured. This was done by first removing the stents followed by dilation of the tract with a radial expansion balloon and insertion of a forward viewing gastroscope through the tract for DEN
  Interventions: Procedure: endoscopic ultrasound; Device: double-pigtail plastic stents

INTERVENTIONS:
Procedure: endoscopic ultrasound — All patients were implanted with stents（DPPS or LAMS）under the EUS
Device: lumen-apposing metal stent — In the LAMS group, patients were stented with LAMS
  Arms: LAMS group
Device: double-pigtail plastic stents — In the DPPS group, patients were stented with DPPS
  Arms: DPPS group

SUMMARY:
Walled-off necrosis (WON) is defined as an encapsulated collection of solid and liquid necrotic material that is usually formed 4 weeks after an episode of acute necrotizing pancreatitis. As the advances in endoscopic techniques and accessories, Endoscopic ultrasound (EUS)-guided transluminal drainage has evolved to become the treatment of choice for symptomatic pancreatic walled-off necrosis (WON). This article aims to compare the efficacy and safety of a double mushroom head metal stent and a double pigtail plastic stent in the treatment of encapsulated necrosis of the pancreas.

DETAILED DESCRIPTION:
According to the revised Atlanta classification, pancreatic fluid collections (PFCs) include acute peripancreatic fluid collections(APFCs) and acute necrotic collections(ANCs), which, over time, turn into pancreatic pseudocysts (PPs) and walled-off pancreatic necrosis (WON). Drainage of these PP and WON is required when they increase in size and become infected or become symptomatic.

Traditionally, WON has been managed surgically, however, surgical necrosectomy is associated with substantial morbidity and mortality, particularly when pursued early. In recent years, with the development of minimally invasive techniques, Endoscopic ultrasound (EUS)-guided transluminal drainage has evolved to become the treatment of choice for symptomatic pancreatic walled-off necrosis (WON).

Double-pigtail plastic stents(DPPS) is the earliest stent used for WON drainage in ultrasound endoscopy, however, These stents are limited by their small diameter leading to increased risk of stent obstruction. Recently, lumen-apposing metal stents (LAMS) have been increasingly used because of the advantage of better lumen apposition and wider diameter, improving access for endoscopic debridement. However, more adverse events(AEs) such as bleeding have been reported.

This article aims to compare the efficacy and safety of DPPS and LAMS in the treatment of Walled-off necrosis

ELIGIBILITY:
Inclusion Criteria:

* Obtention of a written informed consent
* According to Revised Atlanta Classification, abdominal CT/MRI and EUS were diagnosed as WON
* The diameter of WON ≥6cm
* Patient capable of fill in the quality of life questionnaire
* The distance between the EUS-probe and WON was < 1 cm.

Exclusion Criteria:

* No written informed consent
* pancreatic cystic tumor, pancreatic cancer and other benign and malignant tumors
* pancreatic pseudocyst
* WON too far from the stomach and duodenum to perform endoscopic drainage
* Serious abnormalities in liver and kidney function and coagulation function
* Pregnant, parturient or breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
clinical success (clinical improvement and resolution of WON) | two months
  compare rates of WON resolution in patients with LAMS and DPPS for treatment of walled-off necrosis

SECONDARY OUTCOMES:
Adverse Events | two months
  Number of participants with adverse events; type, frequency and intensity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhang, M.S, Study Director — First People's Hospital of Hangzhou
Locations (1):
- Jianfeng Yang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No